CLINICAL TRIAL: NCT04968886
Title: Multicenter Prospective Evaluation of Rapid Viability Tests for Mycobacterium Tuberculosis to Improve the Follow-up of Tuberculosis Patients and Guide Isolation Measures
Brief Title: TuBerculosis Viability Interregional Study and Agreement on Biological Tests
Acronym: TBVISA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180578
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Hospital infection control; Isolation; Treatment response; Tuberculosis; Viability stain
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: viability test on sputum and comparision with culture results (reference test) — Diagnostic Test: viability test on sputum and comparision with culture results (reference test)

SUMMARY:
The objective of the present study is to confirm in a multicentric study the utility of our viability test in large cohort of smear-positive pulmonary tuberculosis patients under treatment and to determine if the test could help physicians to discontinue isolation measures in hospital setting.

DETAILED DESCRIPTION:
When patients with pulmonary tuberculosis (TB) are hospitalized for diagnosis and treatment, isolation measures are mandatory in order to prevent transmission. Recommendations are to maintain isolation until patients are no more infectious, which is ascertained when cultures of respiratory specimens become negative (culture conversion). After administration of antibiotics, the average time to culture conversion is one month for patients with drug-susceptible TB, but 5%-30% cases require more than two months and up to 6 months can be required for multiresistant (MDR)-TB.

Microscopic examination of bacilli in respiratory samples is mainly used as a surrogate marker but because bacilli staining does not differentiate alive from dead bacilli, the interpretation of positive smears is misleading. After 1-2 months of treatment, bacilli can be considered dead while they are still alive and isolation measures are thus erroneously discontinued. Conversely, bacilli can be considered viable while they have already been killed by the treatment and patients kept inadequately in isolation.

To overcome the misleading results, attempts have been made to develop viability biomarkers for Mycobacterium tuberculosis (Mtb), the agent of tuberculosis. Studies using RNA or DNA gave convincing results but their cost is not affordable in most part of the world. Those using fluorescein probes are easiest but studies have shown either conflicting results, or have been evaluated only for a short period of time after initiation of therapy.

Thus, we evaluated a fluorescent staining able to differentiate dead bacilli from alive, which was previously used for detection of industrial environmental pathogens - the Live/Dead® BacLight™ Bacterial viability test (Invitrogen, Biocentric, France). Briefly, the test permits to visualize the bacteria using SYTO-9 and propidiumiodide (PI) fluorescent dyes, which both bind to DNA but penetrate specifically cytoplasmic membrane: SYTO-9 penetrates all bacilli, either viable or not, whereas the PI penetrates only in cells with damaged membrane. Consequently, the viable bacteria are impermeable to PI and only fluoresced due to SYTO-9 appearing green under the fluorescent microscope, whereas dead bacteria are marked by both fluorescent dyes and appear red.

We firstly adapted the kit to mycobacteriology and assessed, in in vitro experiments, the concordance of the test with the culture results. Then, we showed in an observational prospective study its accurateness to predict culture results in patients undergoing antituberculous therapy: the viability test correctly predicted all culture-positive samples in the first two months after treatment.

The objective of the present study is to confirm in a multicentric study the utility of our viability test in large cohort of smear-positive pulmonary tuberculosis patients under treatment and to determine if the test could help physicians to discontinue isolation measures in hospital setting.

Since the test is quick (less than 1 h for the test versus a median of 23 days for culture) and easy to perform, it would be useful to help physicians to maintain isolation in clinical settings while avoiding unnecessary cultures. Since the test is also cheap (<1 € for reagents) this issue could be particularly valuable in countries with limited resources and where cultures are unavailable.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 years old
* Patient put on anti-tuberculosis treatment for pulmonary tuberculosis with at least one positive ME
* Information given on the study and the right to oppose

Exclusion Criteria:

* Refusal of participation
* People unable to understand the information, In accordance with article 11218 of the public health code,
* people not affiliated with Health Insurance,
* pregnant or breastfeeding women patients under legal protection can be included in a non-interventional study (type 3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Smear-positive pulmonary tuberculosis patients.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Result of the viability test (positive or negative) compared to culture results (reference test). - The reference test will be considered as positive (C+) if Mtb are grown on solid or liquid media et negative (C-) if the cultures remain sterile after 42 | 12 months
  The culture will be judged positive in case of isolation of tubercle bacilli in solid or liquid medium and will be judged negative if the culture is sterile after 42 days of incubation in liquid medium and 60 days in solid medium. If the culture is contaminated with bacteria other than tubercle bacilli, it will be considered uninterpretable.
  - The microscopic viability test will be judged positive in the event of observation of at least 1 bacillus per slide is stained with Syto9 in fluorescent green per slide on microscopic examination of the smear and will be judged negative if no bacillus fluoresces in green .
  Each test will be interpreted blind to the results of the other and the results of the TVmol. the diagnostic indices of the microscopic viability test will be calculated

SECONDARY OUTCOMES:
Evaluate the diagnostic performance of the molecular test for the viability of tuberculosis bacilli | 12 months
  Using real-time Polymerase Chain Reaction amplification in comparison with the bacterial culture (reference test).
Study the correlation between the quantitative results of viability tests and the quantitative results of the culture | 12 months
  Microscopic viability test expressed as the number of fluorescent green bacilli, and culture results expressed in number of colonies for culture in solid medium and Molecular viability test expressed in number of amplification cycles to reach the positivity threshold and in molecular concentration of the target gene and the culture results expressed
Evaluate the potential benefit of viability tests for the patient and the hospital over the duration of isolation and the time to discharge from hospital | 12 months
  Evaluate the potential benefit of viability tests for the patient and the hospital over the duration of isolation and the time to discharge from hospital
Describe the cohort of patients hospitalized for pulmonary tuberculosis with positive microscopic examination in the 10 participating centers | 12 months
  Describe the cohort of patients hospitalized for pulmonary tuberculosis with positive microscopic examination in the 10 participating centers

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin WYPLOSZ, Ph, Principal Investigator — Public Assistance of Paris Hospitals (APHP)